CLINICAL TRIAL: NCT04424082
Title: Influence of External Dead Space on Volumetric Capnography Derived Parameters in Mechanically Ventilated COVID-19 Patients
Brief Title: External Dead Space in Ventilated COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Jacob Karlsson, MD PhD, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Karolinska
Record Dates: First submitted 2020-06-07; First posted 2020-06-09 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Coronavirus; ARDS, Human
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dead space removal (Other): external dead space will be removed and Vcap parameters (VCO2, PaCO2 and alveolar dead space) recorded before and after.
  Interventions: Other: Removal of dead space filter

INTERVENTIONS:
Other: Removal of dead space filter — Dead space filters will be removed and Vcap parameters (VCO2 ml/min, PaCO2 kPa, alveolar dead space in ml) recorded before and after removal

SUMMARY:
The objective is to investigate the efficacy of volumetric capnography to detect changes in dead space, CO2 elimination and shape factor parameters before and after disconnection of external dead space in ventilated COVID-19 patients.

DETAILED DESCRIPTION:
Covid-19 patients under mechanical ventilation are currently managed with a lung protective strategy derived from ARDSnet recommendations. In order to minimize the risk of spread of coronavirus, filters and associated respiratory tubing are incorporated to the breathing circuit, thus increasing apparatus dead space with subsequent increase in dead space ventilation. Considering the already often compromised ability for these patients to adequately clear carbon dioxide (VCO2), adding an external dead space can potentially have a substantial impact on CO2 homeostasis. The study will use volumetric capnography (Vcap) to investigate the influence of external dead space on VCO2 and calculated alveolar dead space.

Objective: 1) To investigate the efficacy of Vcap to detect changes in dead space, VCO2 and shape factor parameters before and after disconnection of external dead space.

2) To register the external dead space impact on arterial carbon dioxide tension (PaCO2).

3) To calculate the alveolar dead space based on Vcap data and arterial blood gas analysis results.

Design and setting: Prospective observational study in an intensive care center for Covid-19 patients in a university hospital.

Patients: Covid-19 positive patients of all age groups under mechanical ventilation. Exclusion criteria is ongoing ECMO treatment

Measurements and results: Vcap and Tcap parameters will be registered during mechanical ventilation and correlated to an arterial blood gas sample. Part of the apparatus dead space will then be reduced via removal of the heat and moister exchange filter (HME) with added tubing resulting in a reduction in volume of approximately 80 ml (i.e. the known volume of the HME filter and associated tubing). After the apparatus dead space is removed, the Vcap will be recorded for approximately 15 minutes and an arterial blood gas will be drawn at the end of the period. The HME and associated tubing will then be reattached to the breathing circuit and Vcap and Tcap parameters will be recorded for approximately 30 minutes and an arterial blood gas will be drawn. Vcap data will be analyzed for dead space, slope of phase III, VCO2 and associated shape factor parameters and compared with Tcap parameters. Changes in Vcap parameters will be tested for statistical significance using one and two-way ANOVA for repeated measures and Bland-Altman analysis will be used for comparison.

ELIGIBILITY:
Inclusion Criteria:

Covid-19 positive patients of all age groups under mechanical ventilation

-

Exclusion Criteria:

* Exclusion criteria is ongoing ECMO treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
change in carbon dioxide elimination (VCO2) i.e. ml CO2 eliminated/minute | 60 minutes
  VCO2 is expected to increase after removal of the external dead space

SECONDARY OUTCOMES:
Changes in alveolar dead space (a Vcap derived parameter) | 60 minutes
  Removing the external dead space is expected to decrease alveolar dead space (ml)
Changes in arterial carbon dioxide tension (PaCO2). | 60 minutes
  Removal of external dead space is expected to decrease PaCO2 (kPa).

CONTACTS AND LOCATIONS:
Overall Officials: Björn Persson, MD PhD, Study Director — Karolinska University
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No